CLINICAL TRIAL: NCT05447429
Title: The Effects of Laparoscopic Guided Transversus Abdominis Plane (TAP) Block in Sleeve Gastrectomy Procedure: A Randomized Single Blinded Placebo Controlled Trial
Brief Title: The Effects of Laparoscopic Guided Transversus Abdominis Plane (TAP) Block in Sleeve Gastrectomy Procedure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Sonmez Ocak, Sonmez Ocak,MD, Chief of residents, Samsun Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020.7.2
Record Dates: First submitted 2022-06-25; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Obesity, Morbid; Postoperative Pain; Postoperative Nausea and Vomiting
Keywords: Sleeve gastrectomy; Transversus abdominis plane block; Postoperative pain management
MeSH Terms: conditions — Obesity, Morbid; Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Forty patients had divided into two groups; TAP block group (TAP-B) and placebo (P) group. Every group contained 20 patients and randomization was performed by sealed envelope method. Patient and the data collector resident didn't know the which procedure was done thus single-blinded randomization were provided.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block (Experimental): In this group ,TAP block will be performed with 0.5% 15 ml bupivacaine + 5 ml .
  Interventions: Procedure: Transversus abdominis plane block
- Placebo (Placebo Comparator): In this group , 20 ml saline solution will injected into the transversus abdominis plane.
  Interventions: Drug: Placebo

INTERVENTIONS:
Procedure: Transversus abdominis plane block — TAP block will be performed by a needle which is punctured at the midaxillary line between subcostal margin and iliac crest, once tip of the needle had detected just above the peritoneum the syringe pulled back.
  Arms: TAP Block
Drug: Placebo — 20 ml saline solution will be injected by a needle which is punctured at the midaxillary line between subcostal margin and iliac crest, once tip of the needle had detected just above the peritoneum the syringe pulled back.
  Arms: Placebo

SUMMARY:
Sleeve gastrectomy is the most performed bariatric procedure worldwide. Postoperative pain management is a challenging issue. In this trial, the investigators aimed to explore the effects of laparoscopic guided transversus abdominis plane (TAP) block on postoperative pain management in patient those were performed laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
TAP block is a regional anesthesia technique which could be performed easily especially by laparoscopy and are used in various surgical procedures. In that technique, blockade of the plane between internal oblique muscle and transversus abdominis muscle is performed by infiltration of local anesthesics drugs. Therefore , reduction of postoperative pain could be lead to decrease in postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* patients between 18-65
* undergo Laparoscopic sleeve gastrectomy

Exclusion Criteria:

* Bupivacaine allergy
* having chronic pain or taking pain management
* ASA ( The American Society of Anesthesiologists Physical Classification System) Class 4 or
* Patients who were performed additional procedures including cholecystectomy, hiatal hernia repair or abdominal hernia repair

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) scores | 24th ours
  VAS scores of the patients within 24 hours postoperatively minimun:0 maximum:10
postoperative analgesia doses | within 24 hours postoperatively
  totally consumed analgesics

SECONDARY OUTCOMES:
Nausea and vomiting score | within 24 hours postoperatively
  PONV (Postoperative nausea and vomiting) score calculated with PONV scale: score 0: no nausea or vomiting, score 1:mild nausea, not requesting medication, score 2: moderate nausea requesting medication, score 3: severe nausea and/or vomiting minimum:0 maximum:3
first mobilization and flatus time | within 24 hours postoperatively
  first mobilization and flatus time
time of first opioid administration | within 24 hours postoperatively
  time of first opioid administration

OTHER OUTCOMES:
operation time | time from first incision to last suture
  operation time

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun Research and Training Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coskun M, Yardimci S, Arslantas MK, Altun GT, Uprak TK, Kara YB, Cingi A. Subcostal Transversus Abdominis Plane Block for Laparoscopic Sleeve Gastrectomy, Is It Worth the Time? Obes Surg. 2019 Oct;29(10):3188-3194. doi: 10.1007/s11695-019-03984-4. PMID 31175560
- [Result] Wong KA, Cabrera AG, Argiroff AL, Pechman DM, Parides MK, Vazzana JT, Moran-Atkin EM, Choi JJ, Camacho DR. Transversus abdominis plane block with liposomal bupivacaine and its effect on opiate use after weight loss surgery: a randomized controlled trial. Surg Obes Relat Dis. 2020 Jul;16(7):886-893. doi: 10.1016/j.soard.2020.03.031. Epub 2020 Apr 10. PMID 32402732
- [Result] Saber AA, Lee YC, Chandrasekaran A, Olivia N, Asarian A, Al-Ayoubi S, DiGregorio R. Efficacy of transversus abdominis plane (TAP) block in pain management after laparoscopic sleeve gastrectomy (LSG): A double-blind randomized controlled trial. Am J Surg. 2019 Jan;217(1):126-132. doi: 10.1016/j.amjsurg.2018.07.010. Epub 2018 Aug 1. PMID 30170687
- [Result] Mittal T, Dey A, Siddhartha R, Nali A, Sharma B, Malik V. Efficacy of ultrasound-guided transversus abdominis plane (TAP) block for postoperative analgesia in laparoscopic gastric sleeve resection: a randomized single blinded case control study. Surg Endosc. 2018 Dec;32(12):4985-4989. doi: 10.1007/s00464-018-6261-6. Epub 2018 Jun 4. PMID 29869078